CLINICAL TRIAL: NCT06654440
Title: An Open-label, Multicenter Phase II Clinical Study of SHR-A2102 for Injection in the Treatment of Advanced Gynaecological Malignancies
Brief Title: A Trial of SHR-A2102 for Treatment of Advanced Gynecological Malignancy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-208
Record Dates: First submitted 2024-10-17; First posted 2024-10-23 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-10

CONDITIONS: Advanced Gynecological Malignancy
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental)
  Interventions: Drug: SHR-A2102 for injection

INTERVENTIONS:
Drug: SHR-A2102 for injection — SHR-A2102 for injection

SUMMARY:
The main objective of this study is to evaluate the effectiveness and safety of SHR-A2102 for participants with advanced gynaecological cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Participate in the study voluntarily, sign the informed consent form.
2. Recurrent or metastatic gynecological malignancies that had failed standard treatments.
3. At least one measurable lesion (RECIST version 1.1).
4. ECOG 0~ 1.
5. With adequate organ functions.
6. Female participants of childbearing potential must agree to use highly effective contraception during the treatment period and for at least 7 months after the last dose of SHR-A2102，Female participants' HCG must be negative within 72 hours prior to enrollment and must be non-lactating.

Exclusion Criteria

1. With untreated brain metastasis or concomitant meningeal metastasis and spinal cord compression.
2. Previous or contemporaneous malignancies, unless these malignancies reached complete remission at least 5 years prior before screening and did not require or are not expected to require other treatment during the study period. Such as Cutaneous squamous cell carcinoma, cervical carcinoma in situ etc.
3. Had previously received antibody drug conjugates containing topoisomerase I inhibitors.
4. Had undergone major surgery other than a diagnosis or biopsy within 28 days prior to the first administration; undergone minor traumatic surgery within 7 days prior to first administration.
5. Known to be human immunodeficiency virus positive, active hepatitis B virus, or active hepatitis C virus.
6. Had active pulmonary tuberculosis within 1 year prior to enrolment.
7. Known to be allergic to any of the components of SHR-A2102.
8. Were not fit to participate in this study by investigator's judgment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Radiological scans performed at baseline then every 6 weeks up to 36 weeks, then every 9 weeks thereafter,up to approximately 24 months.
  Assessed by Investigator according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Duration of response (DoR) | Radiological scans performed at baseline then every 6 weeks up to 36 weeks, then every 9 weeks thereafter,up to approximately 24 months.
  Assessed by Investigator according to RECIST 1.1 criteria.
Disease control rate (DCR) | Radiological scans performed at baseline then every 6 weeks up to 36 weeks, then every 9 weeks thereafter,up to approximately 24 months.
  Assessed by Investigator according to RECIST 1.1 criteria.
Time to response (TTR) | Radiological scans performed at baseline then every 6 weeks up to 36 weeks, then every 9 weeks thereafter,up to approximately 24 months.
  Assessed by Investigator according to RECIST 1.1 criteria.
Progression free survival (PFS) | Radiological scans performed at baseline then every 6 weeks up to 36 weeks, then every 9 weeks thereafter,up to approximately 24 months.
  Assessed by Investigator according to RECIST 1.1 criteria.
Overall survival (OS) | follow up once every 60 days. Up to approximately 36 months.
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up.
12 month survival rate | follow up once every 60 days. Up to approximately 24 months.
  Survival rate within one year.
Adverse Events (AEs) | Up to approximately 24 months.
  Include incidence,grade(judged according to NCI-CTCAE V5.0 standards).
PK traits of SHR-A2102: Plasma concentrations of SHR-A2102. | Up to approximately 24 months.
PK traits of SHR-A2102: Plasma concentrations of SHR-A2102 metabolites. | Up to approximately 24 months.
ADA traits of SHR-A2102: Serum concentrations of SHR-A2102 at each planned blood collection time point. | Up to approximately 24 months.
Nab traits of SHR-A2102: Serum concentrations of SHR-A2102 at each planned blood collection time point. | Up to approximately 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided